CLINICAL TRIAL: NCT06979414
Title: Nurse-Led Transfer Programme With Patient Relatives: The Effect of Reducing Transfer Anxiety in Cardiovascular Surgery ICU Patients
Brief Title: Nurse-Led Transfer Program With Family Involvement to Reduce ICU Patient Anxiety
Acronym: FICARE-TX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yakup Akyüz (Other)
Responsible Party: Sponsor-Investigator, Yakup Akyüz, Research Assistant, Department of Surgical Nursing, Istanbul University
Organization: Istanbul University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: İstanbulU/2025/2
Record Dates: First submitted 2025-04-21; First posted 2025-05-19 (Actual); Last update posted 2025-05-19 (Actual); Status verified 2025-04

CONDITIONS: Transfer Anxiety; Intensive Care Unit Discharge; Cardiac Surgery Recovery; Postoperative Anxiety; Critical Care Transition
Keywords: transfer anxiety; patient transfer; intensive care nursing

STUDY DESIGN:
Intervention Model Description: This study was designed as a monocentric, quasi-experimental, parallel-group trial. Participants were assigned sequentially to either the control group or the intervention group based on admission order, without randomization. The intervention group received a structured nurse-led transfer program involving patient relatives, while the control group underwent standard hospital transfer procedures without family involvement. Anxiety levels and vital signs were measured at three time points across both groups for comparison.
Masking Description: No parties were masked in this study due to the nature of the intervention, which involved the visible participation of patient relatives during the ICU transfer process. The open-label design was necessary to ensure ethical and logistical feasibility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-led Transfer With Family Involvement (Experimental): Patients in this group received a structured, nurse-led transfer program involving their primary caregiver. The intervention consisted of three phases: (1) pre-transfer emotional support through a brief ICU visit by the caregiver, (2) accompanied transfer to the general ward led by a nurse and support staff, and (3) post-transfer monitoring of anxiety and vital signs within 30-60 minutes of arrival.
  Interventions: Behavioral: Nurse-led Transfer Programme with Family Involvement
- Standard Transfer Without Family Involvement (No Intervention): Patients in this group underwent the hospital's routine transfer process, which did not include caregiver involvement. Transfers were performed by the ICU nurse and support staff. Anxiety and vital signs were measured at the same three time points as the intervention group: before transfer, immediately prior to transfer, and 30-60 minutes post-transfer.

INTERVENTIONS:
Behavioral: Nurse-led Transfer Programme with Family Involvement — This behavioral intervention was structured in three phases: (1) Pre-transfer preparation, where the patient's primary caregiver visited the ICU for emotional support following verbal instruction and infection control measures; (2) Accompanied transfer to the general ward, led by an ICU nurse, with the caregiver present to provide emotional reassurance; (3) Post-transfer monitoring, where the patient's vital signs and anxiety levels were reassessed within 30-60 minutes of arrival. The goal of the intervention was to reduce ICU transfer-related anxiety through nurse-led, family-involved emotional support.
  Other Names: Family-Inclusive Nurse-led Transfer Program
  Arms: Nurse-led Transfer With Family Involvement

SUMMARY:
This study aims to evaluate whether including a patient's family member during transfer from the intensive care unit (ICU) to the general ward can help reduce anxiety in patients who have undergone cardiovascular surgery. The research is being conducted in a cardiovascular ICU in Turkey. Patients in the intervention group are accompanied by a close relative during the transfer process. Their anxiety levels and vital signs are measured before and after the transfer and compared to those of patients transferred without a relative.

DETAILED DESCRIPTION:
This quasi-experimental study investigates the effect of a nurse-led transfer program involving patient relatives on transfer-related anxiety and vital signs in cardiovascular surgery ICU patients. The study is conducted in a cardiovascular intensive care unit in Turkey between August and October 2024. A total of 150 patients who undergo open-heart surgery and meet the inclusion criteria are enrolled. Participants are assigned sequentially to either the control or intervention group.

In the intervention group, a structured, nurse-led transfer protocol is applied in three phases: (1) pre-transfer preparation involving the patient's relative, (2) accompanied transfer by a relative and clinical staff, and (3) post-transfer monitoring. The control group receives routine hospital transfer procedures, which do not include family involvement.

The primary outcome is the change in patients' state anxiety, measured at three time points (before, immediately prior, and 30-60 minutes after transfer) using the State Anxiety Inventory (STAI-I). Secondary outcomes include changes in vital signs (blood pressure, pulse, respiratory rate, and oxygen saturation), recorded at the same time points.

The study is designed to contribute to the development of family-centered, nurse-led protocols aimed at improving patient comfort and emotional well-being during ICU-to-ward transfers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Undergoing first-time open-heart surgery (e.g., CABG or valve replacement)
* Glasgow Coma Scale (GCS) score ≥ 14 prior to transfer
* Hemodynamically stable at the time of transfer
* Stayed in the cardiovascular surgery ICU for at least 24 hours
* Experiencing first intra-hospital transfer
* Presence of a primary caregiver available for transfer support

Exclusion Criteria:

* Emergency cardiac surgery
* Neurological or psychiatric disorders in the patient
* Postoperative complications resulting in prolonged ICU stay
* Emergency intervention required during the transfer
* Known interpersonal conflict between the patient and the caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in State Anxiety Level Using the State-Trait Anxiety Inventory (STAI-I) | 1. DAY
  The State-Trait Anxiety Inventory - State Form (STAI-I) is a 20-item self-report questionnaire that measures situational anxiety levels. Each item is rated on a 4-point Likert scale. The total score ranges from 20 (lowest anxiety) to 80 (highest anxiety). Higher scores indicate a worse outcome, reflecting greater anxiety levels. The assessment will be conducted at three points: (T1) baseline, (T2) immediately pre-transfer, and (T3) 30-60 minutes post-transfer.

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure | 1. DAY
  Systolic blood pressure will be measured at three time points: (T1) baseline (upon ICU discharge decision), (T2) immediately prior to transfer, and (T3) 30-60 minutes after transfer.
Change in Diastolic Blood Pressure | 1. DAY
  Diastolic blood pressure will be measured at three time points: (T1) baseline (upon ICU discharge decision), (T2) immediately prior to transfer, and (T3) 30-60 minutes after transfer.
Change in Pulse Rate | 1. DAY
  Pulse rate will be recorded at three time points: (T1) baseline (upon ICU discharge decision), (T2) immediately prior to transfer, and (T3) 30-60 minutes after transfer.
Change in Respiratory Rate | 1. DAY
  Respiratory rate will be recorded at three time points: (T1) baseline (upon ICU discharge decision), (T2) immediately prior to transfer, and (T3) 30-60 minutes after transfer.
Change in Oxygen Saturation (SpO₂) | 1. DAY
  Peripheral oxygen saturation (SpO₂) will be measured at three time points: (T1) baseline (upon ICU discharge decision), (T2) immediately prior to transfer, and (T3) 30-60 minutes after transfer.
Predictor of Anxiety Reduction | 1. DAY
  Regression analysis will be performed to evaluate the effect of caregiver presence on the change in patients' state anxiety levels.

CONTACTS AND LOCATIONS:
Overall Officials: yakup akyüz, research assistant, Principal Investigator — istanbul university faculty of nursing department of surgical diseases nursing
Locations (1):
- Izmir Bakircay University Cigli Training and Research Hospital, Cardiovascular Intensive Care Unit, Izmir, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the study publication will be shared. This includes demographic data, STAI-I anxiety scores, and vital signs (blood pressure, heart rate, respiratory rate, and oxygen saturation) measured at three time points. Data will be available beginning 6 months after publication and will be accessible to qualified researchers upon reasonable request to the corresponding author. A data-sharing agreement will be required.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting documents will be available beginning 12 months after publication of the primary results and will be accessible for a period of 5 years.
Access Criteria: Qualified researchers affiliated with academic institutions or healthcare organizations will be able to request access to de-identified individual participant data (IPD), including STAI-I scores, vital signs, and demographic information, as well as the study protocol and statistical analysis plan. Access will be granted upon submission of a data use proposal and signing of a data-sharing agreement. Requests should be submitted to the study contact via email and will be reviewed within 30 days.

REFERENCES:
- [Background] Ortahisar BK, Uslu Y. Intra-hospital transfer anxiety of patients in the neurosurgery intensive care unit: A prospective cohort study. Intensive Crit Care Nurs. 2023 Oct;78:103464. doi: 10.1016/j.iccn.2023.103464. Epub 2023 Jun 22. PMID 37354694
- [Background] Ghorbanzadeh K, Ebadi A, Hosseini M, Madah SSB, Khankeh H. Challenges of the patient transition process from the intensive care unit: a qualitative study. Acute Crit Care. 2021 May;36(2):133-142. doi: 10.4266/acc.2020.00626. Epub 2021 Jan 28. PMID 33508186
- [Background] Dziadzko M, Mazard T, Bonhomme M, Raffin M, Pradat P, Forcione JM, Minjard R, Aubrun F. Preoperative Anxiety in the Surgical Transfer and Waiting Area: A Cross-Sectional Mixed Method Study. J Clin Med. 2022 May 9;11(9):2668. doi: 10.3390/jcm11092668. PMID 35566793
- [Background] de Grood C, Leigh JP, Bagshaw SM, Dodek PM, Fowler RA, Forster AJ, Boyd JM, Stelfox HT. Patient, family and provider experiences with transfers from intensive care unit to hospital ward: a multicentre qualitative study. CMAJ. 2018 Jun 4;190(22):E669-E676. doi: 10.1503/cmaj.170588. PMID 29866892
- [Background] Cheng F, Yan H, Zhong J, Yang H, Nan R, Wang X, Wei Z, Dou X. Knowledge, attitude and practice of registered nurses toward ICU patients' transfer anxiety in China: A cross-sectional study. Heliyon. 2024 Apr 5;10(8):e29318. doi: 10.1016/j.heliyon.2024.e29318. eCollection 2024 Apr 30. PMID 38660287
- [Background] Chen Y, Peet J, Murray L, Ramanan M, Jacobs K, Brailsford J, Osmond A, Kajevu M, Garrett P, Tabah A, Mock C, Lin FF. Waiting to be discharged from intensive care units: Key factors shaping patient and family experiences. Intensive Crit Care Nurs. 2025 Apr;87:103961. doi: 10.1016/j.iccn.2025.103961. Epub 2025 Feb 5. PMID 39914326
- [Derived] Akyuz Y, Er S, Bozok S, Uslu Y. Nurse-Led Transfer Programme With Patient Relatives: Effect on Reducing Transfer Anxiety in Intensive Care Unit Patients. Nurs Crit Care. 2025 Sep;30(5):e70153. doi: 10.1111/nicc.70153. PMID 40919712
- See also: Related Info — https://ebcj.mums.ac.ir/article_23311.html